CLINICAL TRIAL: NCT05134948
Title: A Phase 1/2 Study of Relatlimab (Anti-LAG-3 Monoclonal Antibody) and Nivolumab (Anti-PD-1 Monoclonal Antibody) Fixed-dose Combination in Chinese Participants With Advanced Solid Tumors (RELATIVITY 059)
Brief Title: A Study to Assess Relatlimab and Nivolumab Fixed-dose Combination in Chinese Participants With Advanced Solid Tumors
Acronym: RELATIVITY 059
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA224-059
Record Dates: First submitted 2021-11-16; First posted 2021-11-26 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors
Keywords: BMS-986213

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort A: BMS-986213 Fixed Dose Combination (Experimental)
  Interventions: Drug: BMS-986213
- Cohort B: BMS-986213 Fixed Dose Combination (Experimental)
  Interventions: Drug: BMS-986213

INTERVENTIONS:
Drug: BMS-986213 — Specified dose on specified days

SUMMARY:
The purpose of this study is to assess the safety, drug levels, immunogenicity and preliminary efficacy of BMS-986213 (nivolumab-relatlimab fixed-dose combination) in Chinese participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one lesion with measurable disease as defined by RECIST v1.1 criteria for response assessment
* Participants must have received, and then progressed, or been intolerant to at least one standard treatment regimen in the advanced or metastatic setting, if such a therapy exists
* ECOG status of 0 or 1
* Life expectancy of ≥ 12 weeks at the time of informed consent per Investigator assessment

Exclusion Criteria:

* Participants with history of severe and/or life-threatening toxicity related to prior immune therapy (eg, anti-CTLA-4 or anti-PD-1/PD-L1 treatment or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways)
* Participants with an active, known or suspected autoimmune disease
* Participants with primary CNS tumors

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Approximately 3 years
Number of Participants with Immune-mediated Adverse Events (IMAEs) | Approximately 3 years
Number of Participants with Serious Adverse Events (SAEs) | Approximately 3 years
Number of Deaths | Approximately 3 years
Number of Participants with AEs Leading to Discontinuation | Approximately 3 years
Number of Participants with Laboratory Abnormalities | Approximately 3 years
Maximum Observed Plasma Concentration (Cmax) of Relatlimab | Approximately 3 years
Time of Maximum Observed Plasma Concentration (Tmax) of Relatlimab | Approximately 3 years
Trough Observed Plasma Concentration (Ctrough) of Relatlimab | Approximately 3 years
Concentration of Relatlimab at the end of a dosing interval (Ctau) | Approximately 3 years
Average concentration of Relatlimab over a dosing interval (Cavg(TAU)) | Approximately 3 years
Area under the concentration-time curve in one dosing interval (AUC(TAU)) of Relatlimab | Approximately 3 years
Total Body Clearance (CLT) of Relatlimab | Approximately 3 years
Observed Concentration of Relatlimab at End of Infusion (Ceoi) | Approximately 3 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by Investigator | Approximately 3 years
Disease Control Rate (DCR) by RECIST v1.1 by Investigator | Approximately 3 years
Duration of Response (DOR) by RECIST v1.1 by Investigator | Approximately 3 years
Best Overall Response (BOR) by RECIST v1.1 by Investigator | Approximately 3 years
Ctrough of Nivolumab | Approximately 3 years
Ceoi of Nivolumab | Approximately 3 years
Number of Anti-drug Antibodies (ADAs) to Relatlimab | Approximately 3 years
Number of ADAs to Nivolumab | Approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- China (2):
  - Local Institution - 0001, Beijing, Beijing Municipality
  - Local Institution - 0002, Fuzhou, Fujian

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com